CLINICAL TRIAL: NCT05388487
Title: A Phase 1 Open-Label Dose-Escalation Study to Evaluate the Tolerability, DLT, Pharmacokinetics, and Preliminary Efficacy of HF1K16 in Patients With Refractory Solid Tumors
Brief Title: Tolerability and Safety of HF1K16 Injection in Patients With Refractory Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: HighField Biopharmaceuticals Corporation (Industry)
Collaborators: Tigermed Consulting Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HF1K16-101(CN)
Record Dates: First submitted 2022-05-04; First posted 2022-05-24 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Dose escalation cohort 1: HF1K16 given QOD at 45 mg/m² (Experimental): The first dosing group (45 mg/m²) will include a sentinel subject receiving one dose followed by a 7-day safety evaluation interval. Three or more subjects will receive 7 doses of HF1K16 QOD at 45 mg/m2 per cycle of 21 days.
  Interventions: Drug: HF1K16 /Arm 45 mg/m²
- Dose escalation cohort 2: Oral ATRA followed by HF1K16 QOD at 90 mg/m² (Experimental): The second dosing group will receive oral ATRA at 45mg/m², and three days later HF1K16 QOD at 90 mg/m2 for 7 times per cycle of 21 days.
  Interventions: Drug: HF1K16 /Arm 90 mg/m²
- Dose escalation cohort 3: HF1K16 QOD at 120 mg/m² (Experimental): The cohort 3 will receive 7 doses of HF1K16 QOD at 120 mg/m² per cycle of 21 days.
  Interventions: Drug: HF1K16 /Arm 120 mg/m²
- Dose escalation cohort 4: HF1K16 QOD at 160 mg/m² (Experimental): The cohort 4 will receive 7 doses of HF1K16 QOD at 160 mg/m² per cycle of 21 days.
  Interventions: Drug: HF1K16 /Arm 160 mg/m²
- Dose escalation cohort 5: HF1K16 QOD at 120mg or180 mg (Experimental): The cohort 5 will receive 7 doses of HF1K16 QOD at 120 mg or 180mg per cycle of 21 days.
  Interventions: Drug: HF1K16 /Arm 120 mg or 180 mg

INTERVENTIONS:
Drug: HF1K16 /Arm 45 mg/m² — HF1K16 is a liposome suspension containing encapsulated ATRA. Drug concentration is 2mg/ml, and infusion should be completed between 60 minutes and 90 minutes
  Arms: Dose escalation cohort 1: HF1K16 given QOD at 45 mg/m²
Drug: HF1K16 /Arm 90 mg/m² — HF1K16 is a liposome suspension containing encapsulated ATRA. Drug concentration is 2mg/ml, and infusion should be completed between 60 minutes and 90 minutes
  Arms: Dose escalation cohort 2: Oral ATRA followed by HF1K16 QOD at 90 mg/m²
Drug: HF1K16 /Arm 120 mg/m² — HF1K16 is a liposome suspension containing encapsulated ATRA. Drug concentration is 2mg/ml, and infusion should be completed between 60 minutes and 90 minutes
  Arms: Dose escalation cohort 3: HF1K16 QOD at 120 mg/m²
Drug: HF1K16 /Arm 160 mg/m² — HF1K16 is a liposome suspension containing encapsulated ATRA. Drug concentration is 2mg/ml, and infusion should be completed between 60 minutes and 90 minutes
  Arms: Dose escalation cohort 4: HF1K16 QOD at 160 mg/m²
Drug: HF1K16 /Arm 120 mg or 180 mg — HF1K16 is a liposome suspension containing encapsulated ATRA. Drug concentration is 2mg/ml, and infusion should be completed between 60 minutes and 90 minutes
  Arms: Dose escalation cohort 5: HF1K16 QOD at 120mg or180 mg

SUMMARY:
HF1K16 is an investigational pegylated liposome formulation of All-Trans Retinoic Acid (ATRA) for the induction of remission in patients with acute promyelocytic leukemia (APL) and for the treatment of solid tumors through targeting myeloid derived suppressor cells (MDSCs).

DETAILED DESCRIPTION:
Myeloid Derived Suppressor Cells (MDSCs) play important roles in constituting the immune suppressive environment promoting cancer development and progression. While previous studies had shown that all-trans retinoic acid (ATRA) could induce MDSC differentiation and maturation, the very poor solubility and fast metabolism of the drug limited its applications as an immune-modulator for cancer immunotherapy

HF1K16 is an investigational pegylated liposome formulation with great ATRA dose loading capacity and sustained drug release property. In preclinical studies, HF1K16 was shown to be able to remodel the host systemic immune homeostasis as well as modify tumor microenvironment (TME). It promotes MDSCs maturation into DCs and facilitates immune responses against cancer cells.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide the test of informed consent in writing.
2. Male or female, age > 18 years and < = 75 years.
3. The subjects had to be diagnosed by histology and/or cytology with locally advanced or metastatic solid tumor. There is no effective standard of care or the patient is intolerant to the standard therapy.

   Cohort 5: The subjects must be diagnosed with glioma by histology, and the disease has relapsed or progressed after previous treatment, and there is no effective standard treatment or the subject is intolerant to standard treatment.
4. According to the definition of RECIST 1.1, participants must have at least one measurable lesion.

   Cohort 5: at least one lesion that can be measured in two dimensions is required ( RANO criteria).
5. Eastern group (ECOG) tumor physical state to 0 or 1. Cohort 5: According to Karnofsky physical fitness score ≥ 60.
6. Expected lifetime > 12 weeks.
7. Men or women of childbearing age must agree to adopt effective contraception after signing the informed consent form until 180 days after the end of the study. Premenopausal women or those within 2 years after menopause are included.

Exclusion Criteria:

1. Patients received systemic antitumor therapy, including chemotherapy, radiotherapy, biologic therapy, endocrine therapy, or immunotherapy within 3 weeks prior to the first dose, except for the following: Nitrosoureas or mitomycin C within 6 weeks; Oral fluorouracils and small molecule drugs within 2 weeks or within 5 half-life periods of the drug (whichever is longer); Antitumour traditional Chinese medicine within 2 weeks.
2. Adverse effects of previous anti-tumor therapy have not recovered to CTCAE 5.0 grade rating of ≤ grade 1 (except for toxicity judged by the investigator be of no safety risk, such as alopecia, grade 2 peripheral neurotoxicity, etc.)
3. Patients received other unlisted clinical trial drugs or treatments within 28 days prior to the first dose.
4. Taken vitamin A or any vitamin A derivatives within 7 days prior to the first dose.
5. Past history of deep vein thrombosis or pulmonary embolism.
6. Evidence that there is poor control of thyroid diseases, or diseases of the retina.
7. Patients have symptomatic central nervous system (CNS) metastases, meningeal metastases, or a primary CNS tumor that is associated with progressive neurological symptoms. Except that the brain metastases are shown to be stable judged by imaging examination within 4 weeks.

   Cohort 5: The above criteria do not apply to the fifth cohort. The fifth cohort allowed inhaled or topical corticosteroids, or hormone therapy at physiological replacement doses due to adrenal insufficiency; short-term (≤7 days) corticosteroids were allowed for prophylaxis (eg, contrast media allergy) or treatment of non-autoimmune conditions ( For example, delayed-type hypersensitivity reactions caused by exposure to allergens); systemic corticosteroids (≥10 mg/day prednisone, or other equivalent corticosteroids) for 7 consecutive days within 14 days of the first dose are not allowed or Immunosuppressant therapy.
8. Evidences of serious or uncontrolled systemic disease (for example: instability or decompensated respiratory disease, liver or kidney disease)
9. Serious liver and kidney function damage;
10. Has clinical significance of cardiovascular disease;
11. Have known immune inhibitory disease or human immunodeficiency virus (HIV) infection.
12. Patients with severe osteoporosis or with bone metastases with serum 25-hydroxyvitamin D assay values less than 50 nmol/L.
13. Active hepatitis (Hepatitis B: HBsAg-positive and HBV-DNA ≥ 500 cps/mL or 200 IU/mLL; HCV RNA-positive).
14. Persons with known hypersensitivity to any of the active ingredients or excipients or a history of atopic allergic reactions.
15. The pregnancy test positive (blood beta human chorionic gonadotropin - HCG [B] test positive) or lactationWomen.
16. Researchers believe that patients with combined disease may affect the compliance.
17. Participants not willing to or fail to follow the procedure.
18. Cohort 5: Brain MRI not available.
19. Cohort 5: uncontrolled epilepsy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-02-16 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | 30 days after administration
  Defined by the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE V5.0)
Incidence of dose-limiting toxicities(DLT) | 21 days after administration
  Observe the dose limiting toxicity, and Incidence of dose-limiting toxicities(DLT) will be assessed
Respiration rate of Vital Signs by stethoscope | 30 days after administration
  Changes from baseline for respiration rate in breaths per minute of Vital Signs
Red blood cell count in whole blood sample | 30 days after administration
  Changes from baseline for Red blood cell count in whole blood in10^9 /L
Ventricular rate of ECG | 30 days after administration
  Changes from baseline for ventricular rate in beats per minute
Respiration rate in mg μl/h·g of ECG | 30 days after administration
  Changes from baseline for respiration rate in mg μl/h·g
Heart rate in beats per minute in beats per minute of ECG | 30 days after administration
  Changes from baseline for heart rate in beats per minute
Blood pressure by sphygmomanometer | 30 days after administration
  Changes from baseline for blood pressure in mmHg, both systolic and diastolic pressures will be assessed.
Body temperature by thermometer | 30 days after administration
  Changes from baseline for body temperature in Celsius degree
White blood cell count in whole blood sample | 30 days after administration
  Changes from baseline for white blood cell count in whole blood in 10^9 /L
Neutrophil count in whole blood sample | 30 days after administration
  Changes from baseline for neutrophil count in whole blood in 10^9 /L
Hemoglobin concentration in g/dL in whole blood sample | 30 days after administration
  Changes from baseline for hemoglobin concentration in g/dL in whole blood
Prothrombin time in whole blood sample | 30 days after administration
  Changes from baseline for Prothrombin time in s
International standardized ratio in whole blood sample | 30 days after administration
  Changes from baseline for international standardized ratio
International sensitivity index in whole blood sample | 30 days after administration
  Changes from baseline for international sensitivity index
Activated partial thromboplastin time in whole blood sample | 30 days after administration
  Changes from baseline for activated partial thromboplastin time in s
Total bilirubin concentration in whole blood sample | 30 days after administration
  Changes from baseline for total bilirubin concentration in μmol/L
ALT concentration in whole blood sample | 30 days after administration
  Changes from baseline for alanine aminotransferase(ALT) concentration in U/L
AST concentration in whole blood sample | 30 days after administration
  Changes from baseline for aspartate aminotransferase(AST) concentration in U/L
Total protein concentration in whole blood sample | 30 days after administration
  Changes from baseline for total protein concentration in g/L
Urea concentration in whole blood sample | 30 days after administration
  Changes from baseline for urea concentration in mmol/L
Creatinine concentration in whole blood sample | 30 days after administration
  Changes from baseline for creatinine concentration in μmol/L
Total cholesterol concentration in whole blood sample | 30 days after administration
  Changes from baseline for total cholesterol concentration in mmol/L
Triglycerides concentration in whole blood sample | 30 days after administration
  Changes from baseline for triglycerides concentration in mmol/L
HDL-C in whole blood sample | 30 days after administration
  Changes from baseline for high density lipoprotein cholesterol (HDL-C) in mmol/L
LDL-C in whole blood sample | 30 days after administration
  Changes from baseline for low density lipoprotein cholesterol (LDL-C) in mmol/L
PR interval by ECG | 30 days after administration
  Changes from baseline for PR interval in ms of ECG
QRS by ECG | 30 days after administration
  Changes from baseline for QRS in ms of ECG
QT by ECG | 30 days after administration
  Changes from baseline for QT in ms of ECG
QTc by ECG | 30 days after administration
  Changes from baseline for QTc in ms of ECG
Cohort 5: Determination of overall response rate (ORR) according to RANO criteria | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 weeks
  ORR is defined as the proportion of participants with complete response or partial response (CR+PR)
Cohort 5: Duration of response (DOR) | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 weeks
  DOR, defined as the time between the start of the subject's first assessment of CR or PR and the first assessment of PD or death from any cause, according to RANO criteria by the investigator
Cohort 5: disease control rate (DCR) | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 weeks
  DCR , defined as the proportion of subjects with a best overall response of CR, PR, or SD in the study as assessed by the investigator according to RANO criteria
Cohort 5: progression-free survival (PFS). | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 weeks
  PFS, defined as the time between the subject's first dose and the onset of (any aspect of) tumor progression or death from any cause

SECONDARY OUTCOMES:
HF1K16 pharmacokinetic parameters with Cmax | Up to 48 hours postdose
  Maximum plasma concentration (Cmax) after administration of HF1K16
the overall response rate(ORR) of HF1K16 | Once every six weeks in the first year, then once every 12 weeks afterwards through study completion, an average of 1 year
  ORR is defined as the proportion of participants with complete response or partial response (CR+PR)
Peripheral blood mononuclear cells by whole blood sample | Before injection on Day1,7,13, 21 in each cycle（each cycle is 21 days）
  Assessing peripheral blood mononuclear cells after dose in cells/mL
AUC48h by plasma concentration of whole blood sample | Up to 48 hours postdose
  Area under plasma concentration -time curve from 0 time ot 48 h(AUC0-48) after dose
Tmax by plasma concentration of whole blood sample | Up to 48hours postdose
  Peak time (Tmax) after dose
T1/2 by plasma concentration of whole blood sample | Up to 48hours postdose
  Elimination half-life (T1/2) after dose
CL by plasma concentration of whole blood sample | Up to 48 hours postdose
  Clearance (CL) after dose
Vd by plasma concentration of whole blood sample | Up to 48 hours postdose
  Volume of distribution(Vd) after dose
AUClast by plasma concentration of whole blood sample | Up to 48 hours postdose
  Ratios of geometric means of AUClast (Area under the plasma concentration-time curve from zero to time of last quantifiable concentration) after dose
Cohort 5: To assess the changes in MDSC after HF1K16 treatment, including changes in MDSC number | Before injection on Day1 in each cycle（each cycle is 21 days）
  Assessing peripheral blood mononuclear cells after dose in cells/mL
Cohort 5: Incidence of Adverse Events | after administration
  Defined by the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE V5.0)
Cohort 5: To assess the changes in MDSC after HF1K16 treatment, including changes in MDSC phenotype | Before injection on Day1 in each cycle（each cycle is 21 days）
  Assessment of MDSC phenotype in peripheral blood after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Jinsong Wu, MD, Principal Investigator — Huashan Hospital Shanghai
Locations (7):
- China (7):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Xiaoshan Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No